CLINICAL TRIAL: NCT06115941
Title: Using Pre-Operative Incentive Spirometer Reduces Chances of Basal Ateletasis in Patients Undergoing Upper Abdominal Surgeries- A Randomized Control Trial
Brief Title: Using Pre-op Incentive Spirometer Reduces Chances of Basal Atelectasis in Patients Undergoing Upper Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Muhammad Naeem (Other)
Responsible Party: Sponsor-Investigator, Dr. Muhammad Naeem, Head of the Department of Surgery, Pak Emirates Military Hospital
Organization: Pak Emirates Military Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 265
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Cholelithiasis; Epigastric Hernia; Duodenal Perforation
Keywords: Abdominal Surgery; Atelectasis; Incentive spirometry
MeSH Terms: conditions — Cholelithiasis; Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Incentive spirometer group (Experimental): incentive spirometry group" patients were directed to start incentive spirometry, 48 hours prior to surgery. They were given an incentive spirometer and were briefed that they should inhale into the mouth piece of spirometer to lift the balls to the roof of tube and hold for five seconds and then exhale. 13 They were asked to perform 10 such breaths for 6 times in a day till surgery under direct supervision of researcher and this was charted in patient file.
  Interventions: Device: Pre-Op Incentive Spirometer
- No Incentive spirometer group (No Intervention): In group B or "no incentive spirometry group" patients were not asked to perform incentive spirometry.

INTERVENTIONS:
Device: Pre-Op Incentive Spirometer — incentive spirometry group" patients were directed to start incentive spirometry, 48 hours prior to surgery. They were given an incentive spirometer and were briefed that they should inhale into the mouth piece of spirometer to lift the balls to the roof of tube and hold for five seconds and then exhale. 13 They were asked to perform 10 such breaths for 6 times in a day till surgery under direct supervision of researcher and this was charted in patient file.
  Arms: Incentive spirometer group

SUMMARY:
ABSTRACT Objective: To compare frequency of basal atelectasis in patients undergoing upper abdominal surgery who are provided pre-operative incentive spirometry versus those not provided pre-operative incentive spirometry

DETAILED DESCRIPTION:
After patient selection through "non-probability consecutive sampling" Investigator recorded baseline characteristics of our patients including age, gender and body mass index (BMI). Once recorded, patients will be randomly divided into two equal groups (each containing 37 patients). In group A or "incentive spirometry group" patients were directed to start incentive spirometry, 48 hours prior to surgery. They were given an incentive spirometer and were briefed that they should inhale into the mouth piece of spirometer to lift the balls to the roof of tube and hold for five seconds and then exhale. 13 They were asked to perform 10 such breaths for 6 times in a day till surgery under direct supervision of researcher and this was charted in patient file. In group B or "no incentive spirometry group" patients were not asked to perform incentive spirometry.

After this, all the included patients underwent upper abdominal surgery by expert surgical team under general anesthesia. Type of surgery (Laparoscopic Cholecystectomy / Open Cholecystectomy / perforated duodenal repair/ Epigastric Hernia Repair / Gastrojejunostomy) and duration for which patient was on ventilator support (in minutes) was documented. After surgery, all the patients were given adequate analgesia and antibiotics as per standard hospital protocol. Patients were assessed at 48 hours after surgery for presence of basal atelectasis which will be diagnosed clinically by presence of new onset respiratory symptoms "cough, crackles, tachypnea and reduced breath sounds at bases" and by chest X-ray "presence of basal opacification, crowded air bronchograms, crowded pulmonary vasculature and compensatory hyper-expansion of surrounding unaffected lung".

"The statistical package for social sciences (SPSS) version 22 software was used for statistical analysis of the data. Normality of test will be checked using Shapiro-Wilk test which showed that age and BMI were normally distributed while duration of ventilatory support was non-normal data. For qualitative variables frequency and percentages were used, whereas for quantitative data mean ± standard deviation and median (IQR) were used. Qualitative variables (gender, type of surgery and presence of basal atelectasis) were compared between groups with the use of chi-square test. Quantitative variable (age and BMI) were compared between groups using Student t-test while (duration of ventilatory support) were compared between groups using Mann-Whittney U-test. A p-value of ≤ 0.05 was considered significant".

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* Both gender
* ASA I and II
* Upper abdominal surgeries

Exclusion Criteria:

* Lower abdominal surgeries,
* ASA III-V status,
* Co-morbidities [like diabetes (HbA1C% ≥ 6.5% 11), hypertension
* Smoking
* Chronic lung condition (like asthma, chronic obstructive pulmonary disease, emphysema)
* Pulmonary tuberculosis
* Structural deformity of chest.

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Decreased frequency in post operative Basal Atelectasis | 48 hours after surgery
  After surgery, all the patients were given adequate analgesia and antibiotics as per standard hospital protocol. Patients were assessed at 48 hours after surgery for presence of basal atelectasis which will be diagnosed clinically by presence of new onset respiratory symptoms "cough, crackles, tachypnea and reduced breath sounds at bases" and by chest X-ray "presence of basal opacification, crowded air bronchograms, crowded pulmonary vasculature and compensatory hyper-expansion of surrounding unaffected lung

CONTACTS AND LOCATIONS:
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No